CLINICAL TRIAL: NCT02178891
Title: A 5-year Clinical Evaluation on Brånemark System® RP Ø4.5x4.5 mm Implants
Brief Title: Extra Short Implants Brånemark System® RP Ø4.5x4.5 mm Implants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Nobel Biocare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: T-163
Record Dates: First submitted 2014-06-27; First posted 2014-07-01 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Healthy Volunteers With Severely Resorbed Jaws in Need of an Implant Supported Restoration
Keywords: short implants; Nobel Biocare; partially edentulous; maxilla or mandible

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- short implants (Other)
  Interventions: Device: extra short implant

INTERVENTIONS:
Device: extra short implant

SUMMARY:
An extra short, 2-piece implant with a Brånemark hexagon interface was developed with a bone anchoring length of only 4.5 mm, for subjects with severely resorbed jaws.

ELIGIBILITY:
Inclusion Criteria:

* The subject should be at least 18 years of age and have passed secession of growth
* The subject should be in need of an implant-supported restoration in the posterior region of the mouth (maxilla: first premolar to third molar, mandible: first premolar to second molar, not third molar due to mobile gingiva), where at least 2 implants are needed of which at least one should be an Extra Short Implant
* Obtained informed consent from the subject
* The subject must be in such a physical and mental condition that a 5-year follow-up period can be carried out without foreseeable problems
* The subject should have a severely resorbed posterior mandible and/ or maxilla.
* Implants are only to be placed in healed sites, defined as a site with minimum 6 months of healing following tooth extraction
* At least 6 mm residual bone width, between 4-7 mm residual bone height in the maxilla and between 6-9 mm residual bone height in the mandible
* At implant installation the implant should be stable; final tightening torque of the implant about 25 Ncm or higher, preferably not exceeding 45 Ncm
* The subject should be healthy and compliant with good oral hygiene
* Favorable and stable occlusal relationship

Exclusion Criteria:

* The subject is not able to give her/his informed consent of participating
* Health conditions, which do not permit the surgical treatment
* Reason to believe that the treatment might have a negative effect on the subject's total situation (psychiatric problems), as noted in subject records or in subject history
* Any disorders in the planned implant area such as previous tumours, chronic bone disease or previous irradiation
* Alcohol or drug abuse as noted in subject records or in subject history.
* Heavy smoking (>10 cigarettes/day)
* Intake of medication containing bisphosphonates
* Uncontrolled diabetes, i.e. a subject with diagnosed diabetes that has a history of neglecting doctor's recommendations regarding treatment, food and alcohol intake
* Severe bruxism or other destructive habits
* Immediate insertion (i.e. placement of the implant immediately after extraction)
* Bone augmentation procedures before or at implant installation is not allowed
* Deviation from stated drilling protocol, utilizing osteotomes, is not allowed
* Lack of opposing dentition
* Single crown restorations are not to be performed in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2010-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
marginal bone level changes | yearly, up to 5 years

SECONDARY OUTCOMES:
cumulative survival and success rates | yearly, up to 5 years

OTHER OUTCOMES:
difference between maxilla and mandible | yearly, up to 5 years

CONTACTS AND LOCATIONS:
Locations (2):
- Germany (2):
  - Universtätsmedizin Mainz, Mainz, Rhl-Palat.
  - Universitätsmedizin Mainz, Mainz